CLINICAL TRIAL: NCT05709808
Title: The Effect of Kinesio-Taping on Mild Ankle Instability in Recreational Runners
Brief Title: Kinesio-Taping and Ankle Instability in Recreational Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Responsible Party: Principal Investigator, Hisham Mohamed Hussein, Assistant professor, University of Hail
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12911
Record Dates: First submitted 2022-12-10; First posted 2023-02-02 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Ankle Instability
Keywords: ankle instability; recreational runners; postural stability; Kinesio-Taping
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: randomized controlled trials contain 2 groups
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: all components of the study will be concealed to the allocation process. while the participants, investigator (who collect data), and statistician will be blinded till the end of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mixed group (Experimental): This taping technique is designed to guard against lateral ankle sprains. Kinesio-tape will be applied to the unstable ankle for a lateral ankle sprain. 4 strips of the tape with different stretching percentages will be applied while the ankle joint in a relaxed position.
  ankle exercises will be conducted for 8 weeks, 3 times/ week, each session will last for 60 minutes.
  A standard proprioceptive training program will be implemented three times a week. The training includes both static and dynamic balance on Wobble board with the eyes open while the last stage will be repeated with the eyes closed.
  Interventions: Other: Kinesio-taping; Other: exercises; Other: mixed kinesiotape plus exercises
- Exercise group (Active Comparator): received exercises and proprioceptive training similar as described in the experimental group
  Interventions: Other: exercises
- Kinesio-tape group (Experimental): will receive Kinesio-tape only as described in the mixed group This taping technique is designed to guard against lateral ankle sprains. Kinesio-tape will be applied to the unstable ankle for a lateral ankle sprain. 4 strips of tape with different stretching percentages will be applied while the ankle joint in a relaxed position.
  Interventions: Other: Kinesio-taping

INTERVENTIONS:
Other: Kinesio-taping — kinesiotape is a method of taping used to improve support and increase proprioceptive awareness of the joint, while the exercise program was designed to improve postural stability and balance
  Arms: Kinesio-tape group; Mixed group
Other: exercises — A standard proprioceptive training program will be implemented three times a week. The training includes both static and dynamic balance on Wobble board with the eyes open while the last stage will be repeated with the eyes closed.
  Arms: Exercise group; Mixed group
Other: mixed kinesiotape plus exercises — kinesiotape is a method of taping used to improve support and increase proprioceptive awareness of the joint, while the exercise program was designed to improve postural stability and balance. A standard proprioceptive training program will be implemented three times a week. The training includes both static and dynamic balance on Wobble board with the eyes open while the last stage will be repeated with the eyes closed.
  Arms: Mixed group

SUMMARY:
this clinical trial intended to investigate the effect of applying kinesiotaping to an ankle with mild instability in the recreational runners.

the authors hypothesize that kinesiotaping might improve postural stability in those patients and facilitate returning to activity

DETAILED DESCRIPTION:
Running as a recreational sport has been considered a very popular sport that has been practiced by people of both genders and in different age groups. This sport does not need a special place or equipment for practice, this advantage further increased its popularity, as well as, it has a great effect on physical and mental health and decreases the mortality rate by 25-40%. Running is contributing to lowering body fats, reduction of weight, increase of lean body mass, improving resting heart rate, enhancing cardiovascular fitness, and helping in the cessation of smoking.

The incidence of people who practice running as an activity is high in European civilization as it reaches up to 12.5-31% of the population. Recreational runners might be at high risk for running-related injuries as reported 6.3 injuries per 1000 training hours in comparison to 3.4 injuries in the other types of sports activities.

It is worth mentioning that, the prevalence of studies for running-related injuries increases with time. Studies have identified the incidence of injuries extends from 25%-85% in running activities. The ankle joint occupies the second place, after the knee joint, as the most vulnerable joint to injury during running. These numbers indicate the importance of injury prevention and emphasize the methods that help in the reduction of recurrence as it was recorded the average time for recovery is 72 days which means a long period of caseation of all activities and a burden on the economy.

While most of the running-related injuries are either gradually onset or due to overuse, sudden ankle injuries might also occur. One of the most common ankle injuries is the lateral sprains of the sub-talar joint. This injury may lead to trauma to the soft tissues and bony components and consequently affect the function of the injured joint.

Ankle sprain causes a decrease in postural stability and neuromuscular control due to improper somatosensory functioning which is linked to this injury on both sides of the lower limbs either on the affected or non-affected one. postural stability is one of the major functions that depend mainly on the cues originating from proprioceptors. Cutaneous stimulation, especially skin stretching, has been considered as an influential factor in joint proprioception. More accurate joint position sense was reported when the skin was stimulated.

Consequently, any therapeutic intervention which can stimulate skin receptors might have positive effects on the related joint proprioception and may enhance the sensorimotor functioning so it might help lower the risk for ankle injuries.

Kinesio tape (KT) is the application of an adhesive and elastic cotton tape on the skin. This tape is anti-allergic and can be left in place for 3 to 5 days without adverse effects. This therapeutic method has gained increasing interest in the field of rehabilitation and sport. It provides a stretching effect on the skin and may stimulate the cutaneous aspect of the proprioception which in turn may affect the somatosensory function.

A study was conducted with KT on medial tibial stress syndrome which showed a reduction of the loading stress in these patients. This syndrome is usually resulted from repeated microtrauma to the tissues and usually reported in physically active persons as recreation runners. Various studies reported significant improvement in postural control, dynamic, static balance, and improving strength after applying the taping on the participants with ankle instability. Even though, a recently published systematic review reported there is limited scientific evidence regarding the use of KT in the rehabilitation of musculoskeletal injuries.

Exercise is still the best intervention for the treatment of patients with ankle instability as it is designed to stimulate proprioception and decrease the risk of ankle injuries. However, specially designed programs and their preventive effect are still inconclusive and need further research. In addition, there is still controversy in using the KT in the rehabilitation of ankle instability as there was a study that reported no significant improvements in the balance measurements.

Most of the studies are conducted on healthy subjects or athletes but no one takes care of non-athletes who are practicing regular activities as recreational runners, as well as, one of the main components of the prevention of injuries and their recurrence is the building up of awareness especially the increase of the popularity of the taping through different media and the increase of using it during competitive matches. So the purpose of this study is to compare the KT versus special proprioceptive training on the postural stability in recreational runners.

ELIGIBILITY:
Inclusion Criteria:

1. healthy college-age males;
2. participate regularly in running activity (1-3 times /week for the last 6 months);
3. Mild ankle instability (score within 24.5-27) according to Cumberland Ankle Instability Tool (CAIT)

Exclusion Criteria:

1. vestibular system problems; and presence of traumatic brain injury in the last three months;
2. fracture or surgery to lower limb;
3. drugs that affect the balance or vestibular system.

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
postural stability | 4 weeks
  measured by the score gained on the appropriate test on biodex balance system. this test has different difficult levels from 1 - 6 with the highest numbet indicated the easiest level. the Biodex device records the number of errors the patient achieve so the higher the patient record the lower the stability score

SECONDARY OUTCOMES:
star excursion test | 4 weeks
  The test initially encourages the maximal reaching of the opposite leg in eight directions while maintaining loading on a single leg. A tape was used to be stuck on the floor and a protractor to divide the tape into 8 directions with 45° in-between. During the examination the participants shod not touch the floor and maintaining their balance, the test repeated three times and the average was calculated. the hgher the reach distance the better the balance status of the participants

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hail, Ha'il, Ha'il Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
all data will be kept in a safe to keep confidentiality of the patient data